CLINICAL TRIAL: NCT01547962
Title: A Pilot Clinical Trial to Assess the Safety and Efficacy of Gintuit (TM) (Allogeneic Cultured Keratinocytes and Fibroblasts in Bovine Collagen) in Establishing a Functional Zone of Attached Gingiva
Brief Title: A Pilot Clinical Trial of Gintuit (TM)in Establishing a Functional Zone of Attached Gingiva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-PER-001
Record Dates: First submitted 2012-02-28; First posted 2012-03-08 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Split-mouth design: Treatment (Experimental)
  Interventions: Device: Gintuit
- Split-mouth design: Control (Active Comparator)
  Interventions: Other: autologous Free Gingival Graft (FGG)

INTERVENTIONS:
Device: Gintuit — Gintuit is prepared in a "S" fold and trimmed to fit the prepared wound bed, with a standardized width of 5 mm and sutured in place with a 5/0 gut suture.
  Arms: Split-mouth design: Treatment
Other: autologous Free Gingival Graft (FGG) — Autologous FGG harvested from the subject's palate, the width of the FGG will be 5 mm and sutured in place with a 5/0 gut suture.
  Arms: Split-mouth design: Control

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Gintuit compared to a free autogenous graft using donor tissue harvested from the subject's palate in the treatment of subjects who have an insufficient zone of attached gingiva associated with at least two non adjacent teeth. The trial is designed to demonstrate non-inferiority between treatment and control in the change in amount of attached gingiva over the 6 month observation period.

Gintuit will be placed as a graft in one of the deficient zones, and a free autogenous graft will be placed in the other. The grafts will be evaluated clinically to determine the change in the amount of attached gingiva and on at least three subjects, a small biopsy will be taken to allow histologic evaluation and comparison of both grafts.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older at the time of enrollment, and not older than seventy years.
2. Subject has at least two non-adjacent teeth with an insufficient zone of attached gingiva which requires soft tissue grafting. The two selected teeth must be located in contralateral quadrants. (In case of adjacent teeth requiring grafting, only one tooth at each site will act as test or control tooth, but both teeth will get the same treatment).
3. Root coverage is not desired or indicated at the time of grafting.
4. Females of childbearing potential must have a documented negative urine or serum pregnancy test.
5. Subjects must have read, understood and signed an institutional review board (IRB) approved Informed Consent Form.
6. Subjects must be able and willing to follow study procedures and instructions.

Exclusion Criteria:

1. Teeth that have an insufficient zone of attached gingiva that would be best treated using soft tissue grafts, which would attempt to cover the denuded root surface.
2. Subjects with any systemic conditions (i.e., diabetes mellitus, cancer, HIV, bone metabolic diseases) which could compromise wound healing and preclude periodontal surgery.
3. Subjects who are currently receiving or have received within one week prior to study entry, systemic corticosteroids (including inhaled), immunosuppressive agents, radiation therapy, and/or chemotherapy which could compromise wound healing and preclude periodontal surgery.
4. Subjects with the presence of acute infectious lesions in the areas intended for surgery.
5. Subjects who smoke.
6. Teeth requiring treatment are molars.
7. Teeth with axial mobility.
8. Known hypersensitivity to bovine collagen.
9. Subjects enrolled in medical, dental, or any investigational device study for any disease within the past four weeks.
10. Subjects who have received an investigational drug or biological treatment within the three months prior to study enrollment (medical or dental).
11. Subjects previously treated with Gintuit, Dermagraft or any other skin graft at the target site(s).
12. Subjects who, in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Amount of attached gingiva | 6 months
  Change in the amount of attached gingiva

SECONDARY OUTCOMES:
Inflammation | week 1, week 4, month 3 and month 6
  Change from baseline in inflammation score
Color of grafted tissue | 4 weeks, 3 months, 6 months
  Color match of the grafted tissue to the adjacent tissue
Texture of grafted tissue | 4 weeks, 3 months, 6 months
  Texture match of the grafted tissue to the adjacent tissue
Oral muscle pull | 6 months
  Resistance to oral muscle pull
Probing depth | 6 months
  Change in probing depth from baseline
Clinical attachment level (ie, distance from the cemento-enamel junction (CEJ; or another definite chosen landmark) to the base of the sulcus or periodontal pocket) | 6 months
  Change in clinical attachment level (mm) from baseline
Overall Subject Preference | 6 months
  VAS scale subject assessment of each treated site with anchors of "disappointed" and "fully satisfied".
Recession depth | 3 months, 6 months
  Change in recession depth
Keratinized tissue | 3 months, 6 months
  Width of keratinized tissue

CONTACTS AND LOCATIONS:
Locations (1):
- PerioHealth, Houston, Texas, United States

REFERENCES:
- [Result] McGuire MK, Scheyer ET, Nunn ME, Lavin PT. A pilot study to evaluate a tissue-engineered bilayered cell therapy as an alternative to tissue from the palate. J Periodontol. 2008 Oct;79(10):1847-56. doi: 10.1902/jop.2008.080017. PMID 18834238